CLINICAL TRIAL: NCT01534793
Title: Observational Study Evaluating the Quality of Laser Enucleation of the Prostate Using a LUMENIS Laser Device
Brief Title: QUAPELLA (QUAlity of Prostate Enucleation by LUMENIS - Laser)
Acronym: QUAPELLA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K070301 / IC0709; 2008-A-00498-47 (Other: IDRCB)
Record Dates: First submitted 2012-01-25; First posted 2012-02-17 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Quality assessment; Benign Prostatic Hyperplasia; Enucleation of the prostate; LUMENIS; Laser; Learning Curve
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HoLEP: Holmium Laser Enucleation of the Prostate
  Interventions: Procedure: Holmium Laser Enucleation of the Prostate (HoLEP)

INTERVENTIONS:
Procedure: Holmium Laser Enucleation of the Prostate (HoLEP) — Under regional or general anaesthesia Urethroscopy to check the location of the prostatic capsule Enucleation of the prostatic lobes (median if present, then lateral lobes)Hemostasis Morcellation Device : LUMENIS Laser

SUMMARY:
This observational study aims at describing the learning curve of the Holmium Enucleation of the Prostate (HoLEP) technique using a LUMENIS laser device by senior attending urologists.

DETAILED DESCRIPTION:
This is a prospective, multicentre observational study studying the learning curve of the HoLEP procedure, through auto-evaluation of the quality of the surgery by senior attending urologists introducing HoLEP in their current clinical practice. This is a single arm, not comparative study. The primary outcome is the ability of each surgeon to perform 4 HoLEP procedures successfully, according to a pre-defined surgical performance scale [varying from 0 to 5]. To be successful, a procedure must be scored 5/5. Each procedure is evaluated at the end of the surgical act by the surgeon himself. As secondary outcomes, the short term efficacy and safety parameters of the HoLEP technique will be evaluated through the following data prospectively collected:

* I-PSS symptom score (15 days before operation, at 6 and 12 months postoperative)
* I-PSS bother score (15 days before operation, at 1, 6 and 12 months postoperative)
* DAN-PSSsex score (15 days before operation, at 6 and 12 months postoperative)Global sexual satisfaction (15 days before operation, at 6 and 12 months postoperative)
* Quality of life score QoL-Europe (15 days before operation, and at 12 months postoperative)
* Urinary flow rate I-PSS symptom score (15 days before operation, at day 0, and at 1, 6 and 12 months postoperative)
* Postvoid residual volume (15 days before operation, at day 0, and at 1, 6 and 12 months postoperative)
* Ultrasound examination of the prostate (15 days before operation, at 6 and 12 months postoperative)
* PSA blood testing (15 days before operation, at 6 and 12 months postoperative)One month post-operative questionnaire at one month post-operative
* Evaluation of adverse events (the day of operation, at 1, 6 and 12 months postoperative)
* Satisfaction of the intervention (at 1 and 12 months postoperative)
* Pathologic examination of the prostate tissue (at 1 months postoperative)
* Blood levels of sodium, haemoglobin, and haematocrit (15 days before intervention, immediately after intervention,)

Time needed for each step of the procedure:

* prostatic capsule contact
* enucleation of the median lobe
* enucleation of the lateral lobes
* hemostasis
* morcellation Laser data (duration, Joules number number of fibers used, fibre type, morcellator ans nephroscope type)
* Tissue weight
* Irrigation volume
* Need for coagulation with another device
* Adverse events during the procedure
* Type of catheter after surgery
* Duration of the catheterization
* Post-operative irrigation (duration, volume, type)
* Hospital stay. The indications of the surgery are the usual indications for bladder outlet obstruction relief in ta context of low urinary tract symptoms due to benign prostatic hyperplasia, as an alternative to the other level 1
* Grade A recommended surgical techniques. The profile of every surgeon will be recorded in terms of surgical experience with age, number of previous endoscopic prostatic surgical procedures, number of laser procedures.

The study design is scheduled as follows:

* Inclusion visit (between D-25 and D-5 before surgery), for inclusion written informed consent as assessment of baseline data
* Surgical intervention (D0): performed as previously described in the literature, with assessment of perioperative data
* One month visit: one month data
* Six month visit: six months data
* One year visit: one year data Statistical analysis will be conducted under SAS9.2 as descriptive analysis for all data, CUSUM technique for main outcome criterion (Altman et al. Stat Med 1988 7 : 629-637 and modelisation of the learning curve.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients over 50
2. Classification of risk according to the American Society of Anesthesiologists (ASA) score: score 1, 2 or 3
3. Protocol accepted by patient (signed informed consent)
4. Patient presenting low urinary tract symptoms due to benign prostatic hyperplasia, since at least 3 months, with indication of surgical relief of bladder outlet obstruction , with International prostate symptom score (I-PSS)≥ 12 and a bother score ≥ 3, or full bladder retention, drained by a catheter or suprapubic catheter
5. Patient with maximum urinary flow rate ≤ 12mL/s for a voiding volume ≥ 125mLat uroflowmetry, for patients who are not drained
6. Prostate weight between 40 and 80 grams
7. Post void residual volume ≤ 300cc, for patients who are not drained
8. Normal renal function
9. Non suspect digital rectal examination
10. PSA value et blood test £ 4 ng/ml, or negative prostatic biopsies if PSA comprised between 4 and 10 ng/ml for patients with age < 75 and life expectancy > 10 years
11. Patient under oral anticoagulation therapy if a therapeutic switch is possible and validated by both the anaesthesiologist and the prescription of the anticoagulation therapy
12. Patient under under antiplatelet agents if this treatment can be interrupted without replacement therapy 5 days prior to surgery without any increased risk for the patient safety
13. Patient gave informed consent and is not opposed to the use of the data collected during the study for research purpose
14. Patient treated by BPH drugs if the duration and type are known, and if the treatment has been stopped before the intervention (one week before surgery for plants and alpha-blockers, one week for 5-alpha reductase inhibitors)
15. Patients has valid health insurance/coverage.

Exclusion Criteria:

1. Patients with unstable known cardiac or pulmonary disease
2. Patients with severe myasthenia, multiple sclerosis, Parkinson disease with known bladder or urinary sphincter dysfunction.
3. Patient with history of severe pelvic injury having caused severe external urinary sphincter damage.
4. Patient with active urinary tract infection
5. Patient with urinary catheter or a suprapubic catheter for a reason other than acute urinary retention due to benign prostatic hyperplasia or experiencing no need to urinate after an event filling than 300cc
6. Patient with neurogenic disease of the urinary tract
7. Patient with known or suspected malignant lesion of the bladder or the prostate
8. Patient with history of previous prostatic surgery
9. Patient with history of bladder stone, major hematuria, urethral stricture, bladder neck stenosis, bladder disease or diabetes with bladder impairment
10. Patient with a prosthesis or material in the region potentially affected by the surgical procedure.
11. Patient with ano-rectal disease
12. Cases where the surgical indication is decided in an emergency context
13. Patient with predictable incomplete follow-up
14. Patient with coagulation disease or abnormalities not covered by the drugs belonging to the categories cited in inclusion criteria 11 and 12
15. All patient condition that the investigator considers as an exclusion criterion

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting low urinary tract symptoms due to benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the ability of each surgeon to perform 4 HoLEP procedures successfully, according to a pre-defined surgical performance scale [varying from 0 to 5]. | participants will be followed for the duration of the intervention, an expected average of 1 hour
  The primary outcome is the ability of each surgeon to perform 4 HoLEP procedures successfully, according to a pre-defined surgical performance scale [varying from 0 to 5]. To be successful, a procedure must be scored 5/5. Each procedure is evaluated at the end of the surgical act by the surgeon himself.

SECONDARY OUTCOMES:
I-PSS symptom score (15 days before operation, at 6 and 12 months postoperative) | 15 days before operation, at 6 and 12 months postoperative)
I-PSS bother score (15 days before operation, at 1, 6 and 12 months postoperative) | 15 days before operation, at 1, 6 and 12 months postoperative
DAN-PSSsex score (15 days before operation, at 6 and 12 months postoperative) | 15 days before operation, at 6 and 12 months postoperative
Global sexual satisfaction (15 days before operation, at 6 and 12 months postoperative) | 15 days before operation, at 6 and 12 months postoperative
Quality of life score QoL-Europe (15 days before operation, and at 12 months postoperative) | 15 days before operation, and at 12 months postoperative
Urinary flow rate I-PSS symptom score (15 days before operation, at day 0, and at 1, 6 and 12 months postoperative) | 15 days before operation, at day 0, and at 1, 6 and 12 months postoperative
Postvoid residual volume (15 days before operation, at day 0, and at 1, 6 and 12 months postoperative) | 15 days before operation, at day 0, and at 1, 6 and 12 months postoperative
Ultrasound examination of the prostate (15 days before operation, at 6 and 12 months postoperative) | 15 days before operation, at 6 and 12 months postoperative
PSA blood testing (15 days before operation, at 6 and 12 months postoperative) | 15 days before operation, at 6 and 12 months postoperative
One month post-operative questionnaire | at 1 month
Evaluation of adverse events (the day of operation, at 1, 6 and 12 months postoperative) | the day of operation, at 1, 6 and 12 months postoperative
Satisfaction of the intervention (at 1 and 12 months postoperative) | at 1 and 12 months postoperative
Pathologic examination of the prostate tissue | at 1 month postoperative
  Pathologic examination of the prostate tissue (at 1 month postoperative)
Blood levels of sodium, haemoglobin, and haematocrit (15 days before intervention, immediately after intervention,) | 15 days befor intervention, immediately after intervention
Intervention duration | participants will be followed for the duration of the intervention, an expected average of 1 hour
Time needed for each step of the procedure | participants will be followed for the duration of the intervention, an expected average of 1 hour
  Time needed for each step of the procedure:
  * prostatic capsule contact
  * enucleation of the median lobe
  * enucleation of the lateral lobes
  * hemostasis
  * morcellation
Laser data | participants will be followed for the duration of the intervention, an expected average of 1 hour
  Laser data (duration, Joules number number of fibers used, fibre type, morcellator ans nephroscope type)
Tissue weight | participants will be followed for the duration of the intervention, an expected average of 1 hour
Irrigation volume | participants will be followed for the duration of hospital stay, an expected average of 1,5 days
Need for coagulation with another device | participants will be followed for the duration of the intervention, an expected average of 1 hour
Adverse events at the day of operation, at 1, 6,12 months post-operative | the day of operation, at 1, 6,12 months post-operative
Type of catheter at the surgery | participants will be followed for the duration of the intervention, an expected average of 1 hour
Duration of the catheterization | participants will be followed for the duration of hospital stay, an expected average of 1,5 days
Post-operative irrigation (duration, volume, type) | participants will be followed for the duration of hospital stay, an expected average of 1,5 days
Hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1,5 days

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand LUKACS, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Urologie - Hôpital Tenon, Paris, Île-de-France Region, France